CLINICAL TRIAL: NCT05467033
Title: Safety Outcomes Post Kidney Biopsy - Randomized Clinical Evaluation of Efficacy of Desmopressin
Acronym: STOP-BLEED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021/ABM/01/00100
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Kidney Biopsy
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): 0,3ug/kg in 100ml 0,9% NaCl managed as intravenous infusion;
  Interventions: Drug: Desmopressin; Drug: intravenous infusion NaCl
- Placebo comparator (Placebo Comparator): 0,9% NaCl managed as intravenous infusion;
  Interventions: Drug: intravenous infusion NaCl

INTERVENTIONS:
Drug: Desmopressin — desmopressin 0,3ug/kg in 100ml 0,9% NaCl managed as intravenous infusion;
  Other Names: Minirin
  Arms: Experimental
Drug: intravenous infusion NaCl — 0,9% NaCl managed as intravenous infusion
  Other Names: 0,9% NaCl

SUMMARY:
It is a randomized, multicenter, double-blind, placebo controlled, interventional clinical trial that will be conducted in Poland, in about 6 Hospital Nephrology Departments to evaluate the safety and effectiveness of desmopressin on the prevention of bleeding after percutaneous needle kidney biopsy in patients with rare and ultrarare glomerulonephritis.

DETAILED DESCRIPTION:
Glomerulonephritis (GN) are rare diseases which carry a high risk of morbidity and mortality. Very often it is diagnosed in the late stage of a disease. One of the reasons might be the fact of a concern for potential complications which might arise from kidney biopsy which is the only procedure which can confirm a diagnosis of glomerulonephritis. According to the map of health needs for Poland the estimated incidence of glomerulonephritis is 40.6 thousand people per year and approximately 1,250 percutaneous renal biopsy (PRB) are performed annually in the adult population.

There are few other studies which analyse the effect of DDAVP administration on the incidence of post-biopsy bleeding events in patients undergoing ultrasound guided PRB without previous coagulopathy. However, there were controversies regarding the potential side effects of DDAVP22 as the studies included only native kidneys biopsies Therefore, a clinical trial is planned with an adequately statistically powered sample of high-risk patients is planned Patients above 18 years old, already qualified by a nephrologist for a kidney biopsy will be randomized with random permuted blocks method into two equal groups (212 patients each) - in one 0,3 micrograms/kg i.v. of desmopressin (in 100 ml of 0,9% NaCl) will be administered one hour before procedure, in the second placebo only (100 ml of 0,9% NaCl). Kidney biopsy will be performed according to standard procedures by an experienced nephrologist with the use of 16G needles during a standard hospitalization with 48 hours of observation. The investigators will assess minor and major bleeding events occurring in the first 24 hours after the procedure (minor: macroscopic haematuria, clinically silent hematoma on kidney ultrasound performed 24 hours after the procedure, haemoglobin decrease above 20% from baseline; major: blood transfusion, embolization, nephrectomy, death indirectly or directly caused by the procedure) and for safety reasons the occurrence of hyponatremia 24 and 48 hours after kidney biopsy

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Ability to provide Informed Consent
3. Qualification by nephrologist to kidney biopsy in accordance to current standards
4. Initial haemoglobin concentration > 8g/dl and PLT count >100 x103/μL
5. Normal range of APTT and INR
6. Blood pressure control defined as SBP<160 mmHg
7. Permitted antiplatelet/antithrombotic drugs: acetylsalicylic acid and heparin
8. No inflammation at the point of biopsy needle insertion

Exclusion Criteria:

1. Initial sodium concentration <130mmol/l
2. Pregnancy and breastfeeding
3. Anaphylactic shock after desmopressin administration (medical history)
4. Necessity of administration other anti-platelet / anti thrombotic drugs other than acetylsalicylic acid, non-fractionated heparin or low molecular weight heparin
5. Decompensated Heart failure
6. Von Willebrand disease (VWD) type II B
7. As per Investigator opinion a medical situation which may lead to increased intracranial pressure (ICP)
8. Hydronephrosis of the biopsied kidney
9. Usage of any prohibited drug before screening :

   * ASA in dosage > 75mg per day
   * Vitamin K antagonist (VKA)
   * Direct oral anticoagulants (DOAC)
   * Low-molecular-weight heparin (LMWH)
   * Unfractionated heparin (UFH)
   * Except situation when dosage of listed above drugs will be adjusted in accordance to protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding events in 24 hours after the procedure | 24 hours after kidney biopsy
  1. Minor bleeding events: macroscopic hematuria; clinically silent hematoma in ultrasound performed 24h after biopsy, decrease in hemoglobin concentration >20% of baseline.
  2. Major bleeding events: erythrocyte transfusion, embolization, nephrectomy, death related directly or indirectly to bleeding.
Bleeding events in 48 hours after the procedure | 48 hours after kidney biopsy
  1. Minor bleeding events: macroscopic hematuria; clinically silent hematoma in ultrasound performed 24h after biopsy, decrease in hemoglobin concentration >20% of baseline.
  2. Major bleeding events: erythrocyte transfusion, embolization, nephrectomy, death related directly or indirectly to bleeding.

SECONDARY OUTCOMES:
Length of hospitalization | 4 years
  Hospitalization time from kidney biopsy till discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Rydzewska-Rosołowska, Assoc.Prof., Principal Investigator — Second Department of Nephrology and Hypertension with Dialysis Unit
Locations (1):
- II Department of Nephrology and Hypertension, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
All de-identified information will be shared upon asking.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication up to 5 years after.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.